CLINICAL TRIAL: NCT05975528
Title: Effect of Sodium-glucose Cotransporter-2 Inhibitor in Cellular Senescence in Patients With Cardiovascular Diseases or Advanced Type 2 Diabetes
Brief Title: Effect of Sodium-glucose Cotransporter-2 Inhibitor in Cellular Senescence in Patients With Cardiovascular Diseases or Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2022-1483
Record Dates: First submitted 2023-06-13; First posted 2023-08-04 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus; Cellular Senescence; Sodium-Glucose Transporter 2 Inhibitors
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sodium-Glucose Transporter 2 Inhibitors; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2 inhibitor user (Experimental)
  Interventions: Drug: SGLT2 inhibitor
- Glimepiride user (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: SGLT2 inhibitor — For the SGLT2 inhibitor group, total drug adminstration days are 180 days, but non-SGLT2 inhibitor administration period is 3 months, and then changed to the SGLT2 inhibitor another 3 months.
  For the SGLT2 inhibitor group, empagliflozin 10mg or dapagliflozin 10mg once daily is administered.
  Arms: SGLT2 inhibitor user
Drug: Glimepiride — For non-SGLT2 inhibitor (glimepiride) administration period is 3 months, and then changed to the SGLT2 inhibitor another 3 months.
  Arms: Glimepiride user

SUMMARY:
Patients with type 2 diabetes (T2D) are more prevalent with aging-related comorbidities and frailty, which leads to a shorter life expectancy than non-diabetic individuals and that this excess mortality is largely attributable to cardiovascular causes.

Therefore, since diabetes accelerates cellular senescence, attenuating aging process in patients with T2D is expected to reduce progression of comorbidities and eventually increase lifespan.

According to previous studies, sodium-glucose cotransporter 2 (SGLT2) inhibitors have shown increased ketone bodies not only in blood but in various tissues including liver, kidney and colon, which could lead to beneficial effects in metabolic diseases. Especially, β-hydroxybutyrate (βHB) inhibits oxidative stress and reduces insulin resistance, which has a positive effect on preventing cardio-renal-metabolic diseases and aging process in patients with T2D.

In this context, SGLT2 inhibitor can be a promising option to alleviate senescence process in patients with T2D. However, despite the accumulating evidence that support anti-senescent effect of SGLT2 inhibitor in preclinical models, no clinical study has investigated association between SGLT2 inhibitor use and senescence patients with T2D.

Thus, the objective of this study is to determine whether the use of SGLT2 inhibitor is associated with anti-senescent effect in patients with T2D, which may expand the indications of SGLT2 inhibitor other than glycemic control.

DETAILED DESCRIPTION:
<Study design>

* Prospective study : Patients with type 2 diabetes who started antidiabetics for the first time or were taking antidiabetics (metformin-based monotherapy or 2- or 3- agent therapy), requiring additional glycemic control by either SGLT2 inhibitor and non-SGLT2 inhibitor(sulfonylurea) are enrolled in this study.
* Drug administration period: Total 180 days, but non-SGLT2 inhibitor administration period is 3 months, and then changed to the SGLT2 inhibitor another 3 months. Health people are also recruited for comparison with patients with T2D.
* Drug administration: For the SGLT2 inhibitor group, empagliflozin 10mg or dapagliflozin 10mg once daily is administered. For the non-SGLT2 inhibitor group (minimum glimepiride 1mg) was administered depending of the patient's glycemic status and hypoglycemic risk.

  * Glimepiride and gliclazide, both belonging to the sulfonylurea class, can be administered interchangeably.
  * Additionally, medication dosages may be adjusted based on blood glucose and test results, and DPP4 inhibitors may be added according to medical judgment, following the guidelines of the Korean Diabetes Association.

< Study methods>

1. After explaining the contents of the study and obtaining consent during hospitalization or outpatient visit, 20ml of additional whole blood is additionally obtained when blood is collected for routine medical purpose. Also, for those agreed to participate in the study, albuminuria and proteinuria are measured and the remaining specimens (5ml) are stored.
2. Among all patients participating in the study, blood and urine samples should be collected to measure the following parameters in each visit (1~3): fasting glucose, fasting insulin, fasting c-peptide, HbA1c, beta-hydroxybutyrate, free fatty acid-fasting, postprandial 90 min glucose/insulin/c-peptide, BUN, creatinine, eGFR, AST, ALT, ALP, GGT, total bilirubin, total protein, albumin, uric acid, total cholesterol, triglyceride, HDL, LDL, WBC, hemoglobin, hematocrit, platelet, c-reactive protein, urinalysis with microscopy. In addition, the following tests including liver fibroscan (Incorporation of fibroscan conducted up to 3 months before/after registration for reference and use during registration) and body composition tests are conducted to check for diabetic complications.

ELIGIBILITY:
<Inclusion criteria for patients with type 2 diabetes and high risk cardiovascular disease>

1. Patients with type 2 diabetes who meet the diagnostic criteria of standard practice guidelines
2. Age between 50 and 85
3. Patients who signed the consent form
4. Patients who meet at least one of the following as a high-risk group for cardiovascular disease:

1) History of myocardial infarction, within the last 3 months 2) Imaging proven coronary artery disease (2 or more coronary arteries or left main coronary artery disease) 3) History of ischemic or hemorrhagic cerebrovascular disease within the last 3 months 4) Imaging proven obstructive peripheral arterial disease 5) Intima media thickness more than 0.9mm or observed plaque 6) estimated glomerular filtration rate between 30-60 7) BMI more than 25kg/m2 accompanied two or more of the following are present: hypertension, current smoker, imaging proven steatohepatitis, alanine aminotransferase more than 40IU/L

<Inclusion criteria for healthy people>

1. Adults 19 years of age or older who do not meet the diagnostic criteria for metabolic syndrome, diabetes, or hyperlipidemia
2. Patients not taking medications related to diabetes or hyperlipidemia
3. BMI less than 25kg/m2

<Exclusion criteria>

1. Those who are unable to participate in clinical trials due to other researchers' judgment
2. Those who cannot read the consent form
3. Patients who refused to fill out the research participation consent form
4. Breastfeeding or pregnant women
5. Type 1 diabetes
6. adrenal insufficiency, growth hormone deficiency, pituitary disease
7. Patients who have undergone bariatric surgery within the past 2 years or gastrointestinal surgery that can cause chronic malabsorption
8. Patients who have taken anti-obesity drugs within the past month or who have received other treatments that can cause weight changes
9. Patients with blood diseases that can cause hemolysis or abnormal red blood cells
10. Patients with active cancer or undergoing chemotherapy
11. Patients with liver disease and cirrhosis who are taking antiviral drugs
12. Patients with autoimmune disease taking steroids and immunosuppressants
13. Organ transplant patients
14. Taking antibiotics or NSAIDs within the last 2 weeks
15. Patients with acute infections in previous 3 months including COVID-19
16. Previous use of GLP-1 receptor agonist, thiazolidinedione, SGLT2 inhibitor
17. Patients with severe hyperglycemia (HbA1c > 10%)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Cellular senescence markers | Changes from baseline to 3 months after use of SGLT2 inhibitors
  Changes of cellular senescence markers (CD57+CD28- T cell, CD87+ monocyte) between SGLT2 inhibitor users and glimepiride users

SECONDARY OUTCOMES:
Changes of Senescence-associated secretory phenotype | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  SASP (Senescence-associated secretory phenotype) : IL-1/6, TNFa, MCP-1
Changes of biochemistry profiles in blood (10^3/μL) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood WBC count (10^3/μL), Platelet counts (10^3/μL)
Changes of biochemistry profiles in blood (g/dL) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood Hemoglobin (g/dL)
Changes of biochemistry profiles in blood (%) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood Hematocrit (%), HbA1c (%)
Changes of biochemistry profiles in blood (mg/dL) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood Creatinine (mg/dL), Total cholesterol (mg/dL), Triglyceride (mg/dL), HDL-cholesterol (mg/dL), Fasting glucose (mg/dL)
Changes of biochemistry profiles in blood (IU/L) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood AST (IU/L), ALT (IU/L), γ-Glutamyl transferase (IU/L)
Changes of biochemistry profiles in blood (mg/L) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood C-Reactive Protein(mg/L)
Changes of biochemistry profiles in blood (μEq/L) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood Free fatty acid-Fasting (μEq/L)
Changes of biochemistry profiles in blood (μU/mL) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood Fasting Insulin (μU/mL)
Changes of biochemistry profiles in blood (mmol/L) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  - Changes in Biochemistry profiles in blood Beta-hydroxybutyrate (mmol/L)
Changes of body composition using Inbody (kg) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  Changes of body composition using Inbody: Skeletal muscle mass (kg) Body fat mass (kg) Right arm muscle mass (kg) Left arm muscle mass (kg) Trunk muscle mass (kg) Right leg muscle mass (kg) Left leg muscle mass (kg)
Changes of body composition using Inbody (cm) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  Changes of body composition using Inbody: Weight circumference (cm) Hip circumference (cm)
Changes of body composition using Inbody (cm2) | Changes from baseline to 3 months/6 months after use of SGLT2 inhibitors
  Changes of body composition using Inbody: Visceral fat area (cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Yong-ho Lee, Principal Investigator — Department of Internal medicine, Yonsei University College of Medicine
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wen CP, Chang CH, Tsai MK, Lee JH, Lu PJ, Tsai SP, Wen C, Chen CH, Kao CW, Tsao CK, Wu X. Diabetes with early kidney involvement may shorten life expectancy by 16 years. Kidney Int. 2017 Aug;92(2):388-396. doi: 10.1016/j.kint.2017.01.030. Epub 2017 Jun 1. PMID 28577854
- [Background] Emerging Risk Factors Collaboration; Di Angelantonio E, Kaptoge S, Wormser D, Willeit P, Butterworth AS, Bansal N, O'Keeffe LM, Gao P, Wood AM, Burgess S, Freitag DF, Pennells L, Peters SA, Hart CL, Haheim LL, Gillum RF, Nordestgaard BG, Psaty BM, Yeap BB, Knuiman MW, Nietert PJ, Kauhanen J, Salonen JT, Kuller LH, Simons LA, van der Schouw YT, Barrett-Connor E, Selmer R, Crespo CJ, Rodriguez B, Verschuren WM, Salomaa V, Svardsudd K, van der Harst P, Bjorkelund C, Wilhelmsen L, Wallace RB, Brenner H, Amouyel P, Barr EL, Iso H, Onat A, Trevisan M, D'Agostino RB Sr, Cooper C, Kavousi M, Welin L, Roussel R, Hu FB, Sato S, Davidson KW, Howard BV, Leening MJ, Leening M, Rosengren A, Dorr M, Deeg DJ, Kiechl S, Stehouwer CD, Nissinen A, Giampaoli S, Donfrancesco C, Kromhout D, Price JF, Peters A, Meade TW, Casiglia E, Lawlor DA, Gallacher J, Nagel D, Franco OH, Assmann G, Dagenais GR, Jukema JW, Sundstrom J, Woodward M, Brunner EJ, Khaw KT, Wareham NJ, Whitsel EA, Njolstad I, Hedblad B, Wassertheil-Smoller S, Engstrom G, Rosamond WD, Selvin E, Sattar N, Thompson SG, Danesh J. Association of Cardiometabolic Multimorbidity With Mortality. JAMA. 2015 Jul 7;314(1):52-60. doi: 10.1001/jama.2015.7008. PMID 26151266
- [Background] Palmer AK, Gustafson B, Kirkland JL, Smith U. Cellular senescence: at the nexus between ageing and diabetes. Diabetologia. 2019 Oct;62(10):1835-1841. doi: 10.1007/s00125-019-4934-x. Epub 2019 Aug 27. PMID 31451866
- [Background] Palmer AK, Xu M, Zhu Y, Pirtskhalava T, Weivoda MM, Hachfeld CM, Prata LG, van Dijk TH, Verkade E, Casaclang-Verzosa G, Johnson KO, Cubro H, Doornebal EJ, Ogrodnik M, Jurk D, Jensen MD, Chini EN, Miller JD, Matveyenko A, Stout MB, Schafer MJ, White TA, Hickson LJ, Demaria M, Garovic V, Grande J, Arriaga EA, Kuipers F, von Zglinicki T, LeBrasseur NK, Campisi J, Tchkonia T, Kirkland JL. Targeting senescent cells alleviates obesity-induced metabolic dysfunction. Aging Cell. 2019 Jun;18(3):e12950. doi: 10.1111/acel.12950. Epub 2019 Mar 25. PMID 30907060
- [Background] Hickson LJ, Langhi Prata LGP, Bobart SA, Evans TK, Giorgadze N, Hashmi SK, Herrmann SM, Jensen MD, Jia Q, Jordan KL, Kellogg TA, Khosla S, Koerber DM, Lagnado AB, Lawson DK, LeBrasseur NK, Lerman LO, McDonald KM, McKenzie TJ, Passos JF, Pignolo RJ, Pirtskhalava T, Saadiq IM, Schaefer KK, Textor SC, Victorelli SG, Volkman TL, Xue A, Wentworth MA, Wissler Gerdes EO, Zhu Y, Tchkonia T, Kirkland JL. Senolytics decrease senescent cells in humans: Preliminary report from a clinical trial of Dasatinib plus Quercetin in individuals with diabetic kidney disease. EBioMedicine. 2019 Sep;47:446-456. doi: 10.1016/j.ebiom.2019.08.069. Epub 2019 Sep 18. PMID 31542391
- [Background] Kim JH, Lee M, Kim SH, Kim SR, Lee BW, Kang ES, Cha BS, Cho JW, Lee YH. Sodium-glucose cotransporter 2 inhibitors regulate ketone body metabolism via inter-organ crosstalk. Diabetes Obes Metab. 2019 Apr;21(4):801-811. doi: 10.1111/dom.13577. Epub 2018 Dec 4. PMID 30407726
- [Background] Han YM, Ramprasath T, Zou MH. beta-hydroxybutyrate and its metabolic effects on age-associated pathology. Exp Mol Med. 2020 Apr;52(4):548-555. doi: 10.1038/s12276-020-0415-z. Epub 2020 Apr 8. PMID 32269287
- [Background] Cunnane SC, Courchesne-Loyer A, St-Pierre V, Vandenberghe C, Pierotti T, Fortier M, Croteau E, Castellano CA. Can ketones compensate for deteriorating brain glucose uptake during aging? Implications for the risk and treatment of Alzheimer's disease. Ann N Y Acad Sci. 2016 Mar;1367(1):12-20. doi: 10.1111/nyas.12999. Epub 2016 Jan 14. PMID 26766547
- [Background] Sedej S. Ketone bodies to the rescue for an aging heart? Cardiovasc Res. 2018 Jan 1;114(1):e1-e2. doi: 10.1093/cvr/cvx218. No abstract available. PMID 29293913
- [Background] Sebastian-Valverde M, Pasinetti GM. The NLRP3 Inflammasome as a Critical Actor in the Inflammaging Process. Cells. 2020 Jun 26;9(6):1552. doi: 10.3390/cells9061552. PMID 32604771
- [Background] Camell CD, Gunther P, Lee A, Goldberg EL, Spadaro O, Youm YH, Bartke A, Hubbard GB, Ikeno Y, Ruddle NH, Schultze J, Dixit VD. Aging Induces an Nlrp3 Inflammasome-Dependent Expansion of Adipose B Cells That Impairs Metabolic Homeostasis. Cell Metab. 2019 Dec 3;30(6):1024-1039.e6. doi: 10.1016/j.cmet.2019.10.006. Epub 2019 Nov 14. PMID 31735593
- [Background] Kim SR, Lee SG, Kim SH, Kim JH, Choi E, Cho W, Rim JH, Hwang I, Lee CJ, Lee M, Oh CM, Jeon JY, Gee HY, Kim JH, Lee BW, Kang ES, Cha BS, Lee MS, Yu JW, Cho JW, Kim JS, Lee YH. SGLT2 inhibition modulates NLRP3 inflammasome activity via ketones and insulin in diabetes with cardiovascular disease. Nat Commun. 2020 May 1;11(1):2127. doi: 10.1038/s41467-020-15983-6. PMID 32358544
- [Background] Madonna R, Barachini S, Moscato S, Ippolito C, Mattii L, Lenzi C, Balistreri CR, Zucchi R, De Caterina R. Sodium-glucose cotransporter type 2 inhibitors prevent ponatinib-induced endothelial senescence and disfunction: A potential rescue strategy. Vascul Pharmacol. 2022 Feb;142:106949. doi: 10.1016/j.vph.2021.106949. Epub 2021 Nov 26. PMID 34843980
- [Background] Trnovska J, Svoboda P, Pelantova H, Kuzma M, Kratochvilova H, Kasperova BJ, Dvorakova I, Rosolova K, Malinska H, Huttl M, Markova I, Oliyarnyk O, Melcova M, Skop V, Mraz M, Stemberkova-Hubackova S, Haluzik M. Complex Positive Effects of SGLT-2 Inhibitor Empagliflozin in the Liver, Kidney and Adipose Tissue of Hereditary Hypertriglyceridemic Rats: Possible Contribution of Attenuation of Cell Senescence and Oxidative Stress. Int J Mol Sci. 2021 Sep 30;22(19):10606. doi: 10.3390/ijms221910606. PMID 34638943
- [Background] Madonna R, Doria V, Minnucci I, Pucci A, Pierdomenico DS, De Caterina R. Empagliflozin reduces the senescence of cardiac stromal cells and improves cardiac function in a murine model of diabetes. J Cell Mol Med. 2020 Nov;24(21):12331-12340. doi: 10.1111/jcmm.15699. Epub 2020 Sep 17. PMID 32940423
- [Background] Sugizaki T, Zhu S, Guo G, Matsumoto A, Zhao J, Endo M, Horiguchi H, Morinaga J, Tian Z, Kadomatsu T, Miyata K, Itoh H, Oike Y. Treatment of diabetic mice with the SGLT2 inhibitor TA-1887 antagonizes diabetic cachexia and decreases mortality. NPJ Aging Mech Dis. 2017 Sep 8;3:12. doi: 10.1038/s41514-017-0012-0. eCollection 2017. PMID 28900540